CLINICAL TRIAL: NCT03086356
Title: Open Label Phase I Trial in Healthy Chinese Male and Female Volunteers to Investigate Pharmacokinetics and Pharmacodynamics of Idarucizumab to Reverse Dabigatran Anticoagulant Activity
Brief Title: Study to Investigate the Pharmacokinetics (PK) and Pharmacodynamics (PD) of Idarucizumab in Chinese Healthy Male and Female Volunteers Who Had Taken Dabigatran Etexilate and Whose Plasma Concentrations of Dabigatran Were at or Close to Steady State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1321.6
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Dabigatran; idarucizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): Dabigatran etexilate alone (days 1-4) and (days 8-10) and with Idarucizumab (day 11)
  Interventions: Drug: Dabigatran etexilate; Drug: Idarucizumab

INTERVENTIONS:
Drug: Dabigatran etexilate — Days 1-4 and Day 8-11
  Other Names: PRADAXA, PRAZAXA
Drug: Idarucizumab — Day 11
  Other Names: PRAXBIND, Praxbind, Prizbind

SUMMARY:
The primary objective of the trial is to investigate the pharmacokinetics and pharmacodynamics of idarucizumab in Chinese healthy male and female subjects following intravenous administration of idarucizumab followed by idarucizumab with 15 minutes interval when administered at or close to the steady state of dabigatran.

Another objective of this trial is to explore the effect idarucizumab on the PK (pharmacokinetic(s)) and PD (pharmacodynamic) parameters of dabigatran.

ELIGIBILITY:
Inclusion criteria:

* Age >= 18 and Age <= 45 years at screening
* Healthy male and female based upon a complete medical history, including vital signs (Blood Pressure, Pulse Rate, and Body Temperature), 12-lead Electrocardiogram and clinical laboratory tests. Women of childbearing potential must be ready and able to use highly effective methods of birth control per International Committee on Harmonisation M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Body weight >=50 kg with body mass index range >=19.0 and <24.0 kg/m2 at Visit 1.
* Signed and dated written informed consent in accordance with Good Clinical Practice and local legislation prior to admission to the trial.

Exclusion criteria:

* Any finding of the medical examination (including Blood Pressure, Pulse Rate, Body Temperature and Electrocardiogram) is deviating from normal and judged as clinically relevant by the investigator
* Any evidence of a clinically relevant concomitant disease according to investigator's clinical judgement
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients) or immune system disease
* Intake of drugs with a long half-life (> 24 hours) within at least 30 days or less than 10 half-lives of the respective drug prior to first trial drug administration
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/corrected QT (QTc) interval.
* Participation in another trial with investigational drug administration within 60 days prior to first trial drug administration
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking during hospitalization
* Alcohol abuse (consumption of more than 20 g per day: e.g., 1 middle-sized bottles of beer, 1 gou [equivalent to 180 mL] of sake))
* Drug abuse or positive drug screening
* Blood donation (400 mL whole blood donation within 12 weeks, 200 mL whole blood donation or blood component donation within 4 weeks) prior to first trial drug administration
* Intention to perform excessive physical activities within one week prior to first trial drug administration or during the trial
* Any laboratory values outside the reference range that are of clinical relevance according to investigator's clinical judgement
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTcF interval >450 ms)
* A history of additional risk factors for torsades de points (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Positive HIV (human immunodeficiency virus) test result at screening examination
* Positive testing for Hepatitis B Antigen and/or a positive Hepatitis C antibody test result at screening examination
* Subjects considered unsuitable for inclusion by the investigator, e.g. are unable to understand and comply with trial requirements, or have any condition which in the opinion of the investigator would not allow safe participation in the trial.
* Subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until 12 weeks after the trial completion. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female (intra-uterine device with spermicide. hormonal contraceptive since at least 8 weeks)
* History or evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies (e.g. cerebral aneurysm, dissecting aorta, central nervous system (CNS) trauma, retinopathy, nephrolithiasis)
* Abnormal values for prothrombin time (PT), activated partial thromboplastin time (aPTT) and thrombocytes considered by the investigator or one of the co-investigators to be clinically relevant
* Creatinine and estimated glomerular filtration rate (GFR) outside the normal range
* Evidence of proteinuria
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Peking University First Hospital, Beijing, China

REFERENCES:
- [Derived] Wang Z, Zhao X, He P, Chen S, Jiang J, Harada A, Brooks S, Cui Y. Idarucizumab Reverses Dabigatran Anticoagulant Activity in Healthy Chinese Volunteers: A Pharmacokinetics, Pharmacodynamics, and Safety Study. Adv Ther. 2020 Sep;37(9):3916-3928. doi: 10.1007/s12325-020-01439-2. Epub 2020 Jul 20. PMID 32691242
- See also: Related Info — https://clinicaltrials.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre, open-label trial in 1 group of healthy volunteers. The trial included a 2-week treatment period during which the subjects were hospitalised at the trial site and a follow-up period of approximately 3 months.
Pre-assignment Details: Healthy male and female volunteers, aged ≥18 and ≤45 years, body weight
  ≥50 kilograms (kg) with a Body Mass Index (BMI) in the range from ≥19 to <24 kilogram per square meter (kg/m2) were included in the trial.
Groups:
- Dabigatran Etexilate+Idarucizumab: During the first part of the treatment period, dabigatran etexilate was administered alone. All subjects received 220 milligram (mg) dabigatran etexilate (capsule) orally twice daily for 3 days (from Days 1 to 3) and a single 220 mg dose on Day 4. During the second part of the treatment period, after a washout period of 3 days, subjects again received dabigatran etexilate (capsule) orally twice daily for 3 days (from Days 8 to 10) and a single 220 mg dose on Day 11. Idarucizumab (solution for infusion) 2 short infusions of 2.5 grams (g) each, with a 15 minute (min) interval was administered intravenously approximately 2 hours (h) after the last dabigatran etexilate administration.
Period: Overall Study
Arm/Group | Dabigatran Etexilate+Idarucizumab
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who received at least 1 infusion of idarucizumab.
Arm/Group | Dabigatran Etexilate+Idarucizumab
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at the time of informed consent Population: TS
  years | 35.6 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: TS
  Participants
    Female | 6
    Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity is not reported in this trial Population: TS
  Participants
    American Indian or Alaska Native | 0
    Asian | 12
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Concentration of Idarucizumab in Plasma (Cmax)
Description: Cmax, maximum measured concentration of idarucizumab in plasma
Time Frame: -0.017, 0.083, 0.167, 0.317, 0.417, 0.45, 0.583, 0.917, 1.417, 2.083, 3.083, 4.083, 6.083, 10.083, 12.083, 24.083, 48.083, 72.083 hours (h)
Population: Pharmacokinetic set (PKS): The PKS included all subjects of the Treated set (TS) who had at least one Pharmacokinetic (PK) parameter analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles (nmol) per litre (L)
Arm/Group | Dabigatran Etexilate+Idarucizumab
Number analyzed (Participants) | 12
nanomoles (nmol) per litre (L) | 30900 (9.86)

2. Primary Outcome: For Diluted Thrombin Time: Area After Subtraction of Baseline Area From Area Under the Effect Curve Over the Time Interval From 2 - 12 Hours (AUEC Above,2-12) on Day 4 and Day 11
Description: For diluted thrombin time: AUEC above,2-12 (area after subtraction of baseline area from area under the effect curve over the time interval from 2 - 12) on day 4 and day 11.
  The standard deviation (SD) presented is actually the percentage coefficient of variation (CV %)
Time Frame: Day 4 and day 11
Population: Pharmacodynamic set (PDS): The PDS included all subjects in the TS who provided at least one evaluable pre-dose and one on-treatment PD observation after the start of dabigatran administration.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dabigatran Etexilate+Idarucizumab
Number analyzed (Participants) | 12
hours
  Day 4 | 8.23 (32.0)
  Day 11 | 0.118 (140)

3. Secondary Outcome: For Sum Dabigatran: Amount of the Analyte Excreted in Urine at Steady State Over the Time Interval 0-74 Hours (Ae0-74,ss ) on Day 4 and Day 11
Description: For sum dabigatran: Ae0-74,ss (amount of the analyte excreted in urine at steady state over the time interval 0-74) on day 4 and day 11 if feasible.
  As per the protocol, day is counted as "Day 1 = 0:00"
Time Frame: 0-2 h, 2-6 h, 6-10 h, 10-12 h,12-14h, 14-26 h, 26-50 h, 50-74 h after drug administration of dabigatran etexilate on Day 4 and Day 11.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg (microgram)
Arm/Group | Dabigatran Etexilate+Idarucizumab
Number analyzed (Participants) | 12
μg (microgram)
  Day 4 | 11700 (30.0)
  Day 11 | 11000 (41.8)

4. Secondary Outcome: For Unbound Sum Dabigatran: Area Under the Concentration-time Curve of the Dabigatran in Plasma at Steady State Over the Time Interval 2 Hours-12 Hours
Description: For unbound sum dabigatran: AUC 2-12,ss (Area under the concentration-time curve of the dabigatran in plasma at steady state over the time interval 2 hours-12 hours).
  As per the protocol, day is counted as "Day 1 = 0:00".
Time Frame: Day 4: 74h, 74.5h, 75h, 76h, 78h, 80h, 84h; Day 11: 242h, 242.083h, 242.25h, 242.333h 243.333h, 244h, 246h, 248h, 252h
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/ milliliter
Arm/Group | Dabigatran Etexilate+Idarucizumab
Number analyzed (Participants) | 12
nanograms*hours/ milliliter
  Day 4 | 1270 (37.0)
  Day 11 | 11.6 (44.3)

5. Primary Outcome: Area Under the Concentration-time Curve of Idarucizumab in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, area under the concentration-time curve of idarucizumab in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles (nmol)*hours (h) per litre (L)
Arm/Group | Dabigatran Etexilate+Idarucizumab
Number analyzed (Participants) | 12
nanomoles (nmol)*hours (h) per litre (L) | 44200 (10.1)

6. Primary Outcome: Amount of Idarucizumab Eliminated in Urine Over the Time Interval From 0 to 72 Hours (h) (Ae0-72)
Description: Ae0-72, amount of idarucizumab eliminated in urine over the time interval from 0 to 72 h.
  As per the protocol, day is counted as "Day 1 = 0:00"
Time Frame: 0-2 h, 2-6 h, 6-10 h, 10-12 h,12-14h, 14-26 h, 26-50 h, 50-74 h after drug administration of dabigatran etexilate on Day 4
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micromole (μmol)
Arm/Group | Dabigatran Etexilate+Idarucizumab
Number analyzed (Participants) | 12
micromole (μmol) | 35.3 (57.1)

ADVERSE EVENTS:
Time Frame: Adverse events from the first intake of treatment until the end of treatment visit; up to 23 days
Groups:
- Dabigatran Etexilate+Idarucizumab: During the first part of the treatment period, dabigatran etexilate was administered alone. All subjects received 220 milligram (mg) dabigatran etexilate (capsule) orally twice daily for 3 days (from Days 1 to 3) and a single 220 mg dose on Day 4. During the second part of the treatment period, after a washout period of 3 days, subjects again received dabigatran etexilate (capsule) orally twice daily for 3 days (from Days 8 to 10) and a single 220 mg dose on Day 11. Idarucizumab (solution for infusion) 2 short infusions of 2.5 grams (g) each, with a 15 minute (min)interval was administered intravenously approximately 2 hours (h) after the last dabigatran etexilate administration.
Arm/Group | Dabigatran Etexilate+Idarucizumab
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate+Idarucizumab (N=12)
Haematoma (Vascular disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Albumin urine present (Investigations) | 12
Alpha 1 microglobulin increased (Investigations) | 12
Protein urine present (Investigations) | 11
Activated partial thromboplastin time prolonged (Investigations) | 10
Urine electrophoresis abnormal (Investigations) | 10
Prothrombin level decreased (Investigations) | 4
Blood triglycerides increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT03086356/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03086356/SAP_001.pdf